CLINICAL TRIAL: NCT02692404
Title: Labor Pain and Postpartum Behavioral Health Outcomes Study
Acronym: LPPD
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Grace Lim, MD, MS, Associate Professor, University of Pittsburgh
Other Study IDs: PRO15030338
Record Dates: First submitted 2016-02-17; First posted 2016-02-26 (Estimated); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Depression, Postpartum; Pregnancy; Child Development; Pain; Labor Pain
Keywords: Postpartum Depression; Perinatal Depression; Pregnancy; Anesthesia; Obstetric; Pain; Analgesia; Epidural; Midwife; Infant Development; Pain Management
MeSH Terms: conditions — Depression, Postpartum; Pain; Labor Pain; Agnosia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva samples for DNA extraction
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Hospital Birth: Healthy nulliparous participants, planning spontaneous vaginal or induced vaginal delivery, and planning delivery at a hospital woman-care birth center (Magee-Womens Hospital of UPMC) will be consented to participate in the study at their 3rd trimester clinic visit. Participants and their newborns will be followed for a period of 3 months postpartum. They will be planning to utilize labor epidural analgesia for pain control during labor.
- Midwife Center Birth: Healthy nulliparous participants, planning vaginal delivery under the primary care of a nurse midwife (The Midwife Center for Birth and Womens Health, or UPMC-Mercy) will be consented to participate in the study at their 3rd trimester clinic visit. Participants and their newborns will be followed for a period of 3 months postpartum. They will be planning to avoid labor epidural analgesia for pain control during labor.

SUMMARY:
In this pilot prospective longitudinal observational study, women who are pregnant and who will be experiencing childbirth for the first time will be recruited at the third trimester and observed longitudinally for psychiatric and pain characteristics until 3 months postpartum. The primary outcome is postpartum depression, assessed by Edinburgh Postnatal Depression Scale (EPDS). Infants will also be observed for infant development characteristics over time. Women who choose to receive labor epidural analgesia will be observed, as well as women who choose to avoid labor epidural analgesia. At baseline, women will complete baseline surveys as well as a baseline pain sensitivity test (quantitative sensory testing, QST). During labor, they will complete an electronic pain diary delivered by a bedside mobile device. Three postpartum assessments will occur over 3 months to assess maternal depression, other psychosocial variables, and infant development.

DETAILED DESCRIPTION:
Our primary goal in this prospective observational study is to observe laboring women's sensitivity to, and characteristics of, labor pain, for the primary outcome of postpartum depression. Secondary endpoints include parenting self-efficacy, maternal-infant attachment, and infant development. The purpose of this pilot phase is to establish study protocol feasibility, and secondarily to determine trends that will inform future sample size calculations for a larger prospective study.

Our key research questions are:

1. What is the association between perceived intensity and unpleasantness of labor pain and postpartum behavioral health outcomes?
2. Do personality, psychological, and genetic factors associated with depression correlate with differences in labor pain experience?

Our hypothesis is that new mothers who have lower pain intensity and unpleasantness during the labor and delivery period will have a reduced risk for postpartum depression, defined by Edinburgh Postnatal Depression Score (EPDS) score. We secondarily hypothesize that women with lower labor pain intensity and unpleasantness scores will have improved maternal-infant attachment, higher parenting self-efficacy, lower perceived stress, and that their infants will exhibit improved child development.

Methods: Baseline assessments of depression, anxiety, resiliency, perceived social support, pain catastrophising, and quantitative sensory testing (QST) will be undertaken. Baseline saliva samples will be collected for future genetic analysis. Throughout labor, pain will be assessed at high density and frequency by an electronic pain diary (mobile app developed by the study team), delivered at the bedside by a portable electronic device (Android tablet) provided by the study team. Labor variables will be recorded, including number of manual epidural supplemental doses, total dose of local anesthetic delivered, and the outcome of labor. Postpartum assessments will include depression, pain inventory, anxiety, perceived stress, maternal-infant bonding, breastfeeding, child development, and parenting self-efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Nulliparous
* Aged ≥18
* Proficiency in English language
* Planning spontaneous or induced labor and delivery
* Planning to avoid labor epidural analgesia (Midwife Center group)
* Planning to utilize labor epidural analgesia (Magee-Womens Hospital group)
* Receiving perinatal care at Magee-Womens Hospital or at The Midwife Center for Birth and Women's Health
* Available and committed for followup at 3 months

Exclusion Criteria:

* Severe maternal obstetric disease
* Known or suspected severe fetal comorbid disease
* Contraindications to neuraxial anesthesia
* Unable to follow study protocol over 3 months
* Plans for newborn adoption

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy, nulliparous women, aged ≥18, planning spontaneous or induced labor and delivery at term gestation. Women who have risk factors for depression will be included. Risk factors are defined as history of abuse (partner, sexual, domestic, childhood, and substance); history of mental illness; lack of social support; and depression or anxiety. Women will have been and will continue to receive perinatal care at Magee-Womens Hospital or at The Midwife Center for Birth and Women's Health (TMC). A subset of women who receive care at TMC will choose to deliver at UPMC Mercy and will plan to avoid labor epidural analgesia. All women and their infants will be available for followup at 3 months.
Sampling Method: Probability Sample
Enrollment: 199 (Actual)
Dates: Start 2016-01; Primary Completion 2017-08-08 (Actual); Study Completion 2017-09-18 (Actual)

PRIMARY OUTCOMES:
Edinburgh Postnatal Depression Score (EPDS) | Postpartum Week 6

SECONDARY OUTCOMES:
Perceived Stress | Postpartum Day 1 or 2
Brief Pain Inventory | Postpartum Day 1 or 2, 6 weeks, and 3 months
Maternal-Infant Attachment | Postpartum Week 6, and 3 months
Parenting Self-Efficacy | Postpartum Week 6, and 3 months
Child Development | Postpartum Week 6, and 3 months
Edinburgh Postnatal Depression Score (EPDS) | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Grace Lim, MD, Principal Investigator — University of Pittsburgh School of Medicine; Magee-Womens Hospital of UPMC
Locations (2):
- United States (2):
  - Magee Womens Hospital of UPMC, Pittsburgh, Pennsylvania
  - The Midwife Center for Birth and Womens Health, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gross KH, Wells CS, Radigan-Garcia A, Dietz PM. Correlates of self-reports of being very depressed in the months after delivery: results from the Pregnancy Risk Assessment Monitoring System. Matern Child Health J. 2002 Dec;6(4):247-53. doi: 10.1023/a:1021110100339. PMID 12512766
- [Background] Schmidt RM, Wiemann CM, Rickert VI, Smith EO. Moderate to severe depressive symptoms among adolescent mothers followed four years postpartum. J Adolesc Health. 2006 Jun;38(6):712-8. doi: 10.1016/j.jadohealth.2005.05.023. PMID 16730600
- [Background] Centers for Disease Control and Prevention (CDC). Prevalence of self-reported postpartum depressive symptoms--17 states, 2004-2005. MMWR Morb Mortal Wkly Rep. 2008 Apr 11;57(14):361-6. PMID 18401329
- [Background] Pearlstein T, Howard M, Salisbury A, Zlotnick C. Postpartum depression. Am J Obstet Gynecol. 2009 Apr;200(4):357-64. doi: 10.1016/j.ajog.2008.11.033. PMID 19318144
- [Background] Hirst KP, Moutier CY. Postpartum major depression. Am Fam Physician. 2010 Oct 15;82(8):926-33. PMID 20949886
- [Background] Wisner KL, Sit DK, McShea MC, Rizzo DM, Zoretich RA, Hughes CL, Eng HF, Luther JF, Wisniewski SR, Costantino ML, Confer AL, Moses-Kolko EL, Famy CS, Hanusa BH. Onset timing, thoughts of self-harm, and diagnoses in postpartum women with screen-positive depression findings. JAMA Psychiatry. 2013 May;70(5):490-8. doi: 10.1001/jamapsychiatry.2013.87. PMID 23487258
- [Background] Lindahl V, Pearson JL, Colpe L. Prevalence of suicidality during pregnancy and the postpartum. Arch Womens Ment Health. 2005 Jun;8(2):77-87. doi: 10.1007/s00737-005-0080-1. Epub 2005 May 11. PMID 15883651
- [Background] Davalos DB, Yadon CA, Tregellas HC. Untreated prenatal maternal depression and the potential risks to offspring: a review. Arch Womens Ment Health. 2012 Feb;15(1):1-14. doi: 10.1007/s00737-011-0251-1. Epub 2012 Jan 4. PMID 22215285
- [Background] Murray L, Arteche A, Fearon P, Halligan S, Goodyer I, Cooper P. Maternal postnatal depression and the development of depression in offspring up to 16 years of age. J Am Acad Child Adolesc Psychiatry. 2011 May;50(5):460-70. doi: 10.1016/j.jaac.2011.02.001. Epub 2011 Apr 5. PMID 21515195
- [Background] Pearson RM, Evans J, Kounali D, Lewis G, Heron J, Ramchandani PG, O'Connor TG, Stein A. Maternal depression during pregnancy and the postnatal period: risks and possible mechanisms for offspring depression at age 18 years. JAMA Psychiatry. 2013 Dec;70(12):1312-9. doi: 10.1001/jamapsychiatry.2013.2163. PMID 24108418
- [Background] Boudou M, Teissedre F, Walburg V, Chabrol H. [Association between the intensity of childbirth pain and the intensity of postpartum blues]. Encephale. 2007 Oct;33(5):805-10. doi: 10.1016/j.encep.2006.10.002. French. PMID 18357852
- [Background] Eisenach JC, Pan P, Smiley RM, Lavand'homme P, Landau R, Houle TT. Resolution of pain after childbirth. Anesthesiology. 2013 Jan;118(1):143-51. doi: 10.1097/ALN.0b013e318278ccfd. PMID 23249931
- [Background] Ding T, Wang DX, Qu Y, Chen Q, Zhu SN. Epidural labor analgesia is associated with a decreased risk of postpartum depression: a prospective cohort study. Anesth Analg. 2014 Aug;119(2):383-392. doi: 10.1213/ANE.0000000000000107. PMID 24797120
- [Background] Hiltunen P, Raudaskoski T, Ebeling H, Moilanen I. Does pain relief during delivery decrease the risk of postnatal depression? Acta Obstet Gynecol Scand. 2004 Mar;83(3):257-61. doi: 10.1111/j.0001-6349.2004.0302.x. PMID 14995921
- [Background] Wisner KL, Stika CS, Clark CT. Double duty: does epidural labor analgesia reduce both pain and postpartum depression? Anesth Analg. 2014 Aug;119(2):219-221. doi: 10.1213/ANE.0000000000000322. No abstract available. PMID 25046776
- [Background] Eapen V, Dadds M, Barnett B, Kohlhoff J, Khan F, Radom N, Silove DM. Separation anxiety, attachment and inter-personal representations: disentangling the role of oxytocin in the perinatal period. PLoS One. 2014 Sep 17;9(9):e107745. doi: 10.1371/journal.pone.0107745. eCollection 2014. PMID 25229827
- [Background] Dennis CL, McQueen K. The relationship between infant-feeding outcomes and postpartum depression: a qualitative systematic review. Pediatrics. 2009 Apr;123(4):e736-51. doi: 10.1542/peds.2008-1629. PMID 19336362
- [Background] Segal S. Labor epidural analgesia and maternal fever. Anesth Analg. 2010 Dec;111(6):1467-75. doi: 10.1213/ANE.0b013e3181f713d4. Epub 2010 Sep 22. PMID 20861420
- [Background] Yoon BH, Romero R, Park JS, Kim CJ, Kim SH, Choi JH, Han TR. Fetal exposure to an intra-amniotic inflammation and the development of cerebral palsy at the age of three years. Am J Obstet Gynecol. 2000 Mar;182(3):675-81. doi: 10.1067/mob.2000.104207. PMID 10739529
- [Background] Impey L, Greenwood C, MacQuillan K, Reynolds M, Sheil O. Fever in labour and neonatal encephalopathy: a prospective cohort study. BJOG. 2001 Jun;108(6):594-7. doi: 10.1111/j.1471-0528.2001.00145.x. PMID 11426893
- [Background] Impey LW, Greenwood CE, Black RS, Yeh PS, Sheil O, Doyle P. The relationship between intrapartum maternal fever and neonatal acidosis as risk factors for neonatal encephalopathy. Am J Obstet Gynecol. 2008 Jan;198(1):49.e1-6. doi: 10.1016/j.ajog.2007.06.011. PMID 18166304
- [Background] Pinto PR, McIntyre T, Ferrero R, Almeida A, Araujo-Soares V. Risk factors for moderate and severe persistent pain in patients undergoing total knee and hip arthroplasty: a prospective predictive study. PLoS One. 2013 Sep 13;8(9):e73917. doi: 10.1371/journal.pone.0073917. eCollection 2013. PMID 24058502
- [Background] Ravindran D. Chronic postsurgical pain: prevention and management. J Pain Palliat Care Pharmacother. 2014 Mar;28(1):51-3. doi: 10.3109/15360288.2013.879249. Epub 2014 Feb 19. PMID 24552601
- [Background] Quinlan J, Carter K. Acute pain management in patients with persistent pain. Curr Opin Support Palliat Care. 2012 Jun;6(2):188-93. doi: 10.1097/SPC.0b013e3283520fb6. PMID 22406985
- [Background] Pandolfo G, Gugliandolo A, Gangemi C, Arrigo R, Curro M, La Ciura G, Muscatello MR, Bruno A, Zoccali R, Caccamo D. Association of the COMT synonymous polymorphism Leu136Leu and missense variant Val158Met with mood disorders. J Affect Disord. 2015 May 15;177:108-13. doi: 10.1016/j.jad.2015.02.016. Epub 2015 Feb 25. PMID 25766270
- [Background] Cox JL, Holden JM, Sagovsky R. Detection of postnatal depression. Development of the 10-item Edinburgh Postnatal Depression Scale. Br J Psychiatry. 1987 Jun;150:782-6. doi: 10.1192/bjp.150.6.782. PMID 3651732
- [Background] Boudarene M, Legros JJ, Timsit-Berthier M. [Study of the stress response: role of anxiety, cortisol and DHEAs]. Encephale. 2002 Mar-Apr;28(2):139-46. French. PMID 11972140
- [Background] Wemm S, Koone T, Blough ER, Mewaldt S, Bardi M. The role of DHEA in relation to problem solving and academic performance. Biol Psychol. 2010 Sep;85(1):53-61. doi: 10.1016/j.biopsycho.2010.05.003. Epub 2010 May 26. PMID 20562010
- [Background] Shirotsuki K, Izawa S, Sugaya N, Yamada KC, Ogawa N, Ouchi Y, Nagano Y, Nomura S. Salivary cortisol and DHEA reactivity to psychosocial stress in socially anxious males. Int J Psychophysiol. 2009 May;72(2):198-203. doi: 10.1016/j.ijpsycho.2008.12.010. Epub 2008 Dec 24. PMID 19141305
- [Background] Wong CA. The promise of pharmacogenetics in labor analgesia...tantalizing, but not there yet. Int J Obstet Anesth. 2012 Apr;21(2):105-8. doi: 10.1016/j.ijoa.2012.02.003. Epub 2012 Mar 9. No abstract available. PMID 22405670
- [Background] Landau R. Genetic contributions to labor pain and progress. Clin Perinatol. 2013 Sep;40(3):575-87. doi: 10.1016/j.clp.2013.05.014. Epub 2013 Jun 27. PMID 23972758
- [Background] Milman N. Postpartum anemia I: definition, prevalence, causes, and consequences. Ann Hematol. 2011 Nov;90(11):1247-53. doi: 10.1007/s00277-011-1279-z. Epub 2011 Jun 28. PMID 21710167
- [Background] Aubuchon-Endsley NL, Thomas DG, Kennedy TS, Grant SL, Valtr T. Interactive relations among maternal depressive symptomatology, nutrition, and parenting. Women Health. 2012;52(3):197-213. doi: 10.1080/03630242.2012.662933. PMID 22533896